CLINICAL TRIAL: NCT05182788
Title: The Efficacy Evaluation of CHOLESWISE Pressed Candy on Cardiovascular Health, a Single Center, Randomized, Doubld-Blind, Placebo Controlled Study
Brief Title: The Efficacy Evaluation of CHOLESWISE Pressed Candy on Cardiovascular Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2021-KY-24-01
Record Dates: First submitted 2022-01-04; First posted 2022-01-10 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo pressed candy (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo pressed candy
- CHOLESWISE pressed candy (Experimental)
  Interventions: Dietary Supplement: CHOLESWISE pressed candy

INTERVENTIONS:
Dietary Supplement: Placebo pressed candy — consume 2 tablets per day for 8 weeks
  Arms: Placebo pressed candy
Dietary Supplement: CHOLESWISE pressed candy — consume 2 tablets per day for 8 weeks
  Other Names: Natto combined Phyllanthus emblica pressed candy
  Arms: CHOLESWISE pressed candy

SUMMARY:
To assess the efficacy evaluation of CHOLESWISE Pressed Candy on cardiovascular disease risk factors

DETAILED DESCRIPTION:
This is a single center, randomized, double-blind and placebo controlled study. Subjects are informed to consume the samples every day for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 30 years old, no gender limit;
* Patients with high blood pressure (systolic blood pressure> 120 mmHg or diastolic blood pressure> 80 mmHg) or high blood lipids (TC ≥ 5.18 mmol/L or TG ≥ 1.7 mmol/L), and no medication is used;
* Fully understand the purpose, benefits, potential risks and side effects of this research, and can objectively cooperate with doctors to complete the examination and assessment of diseases and physical conditions;
* People who voluntarily agree and sign an informed consent form.

Exclusion Criteria:

* People with a history of dyspepsia would affect the absorption of the test product;
* Any situation that may affect trial process, including difficult-to-control organic disease or infection, unstable angina pectoris, congestive heart failure and other severe disease;
* People with symptomatic and difficult-to-control neurological, mental diseases or mental disorders;
* Pregnant or breast-feeding women or women who have a positive result on a pregnancy test;
* Allergic to the components of the test product;
* Take supplementary foods and health supplements with the same efficacy two weeks before and during the test.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-06-09 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in blood pressure (systolic blood pressure, diastolic blood pressure) | Days 1, 28, and 56
  Blood pressure will be measured at the beginning, 4-week, and 8-week time points.
Change from baseline in blood lipid (total-Cholesterol, triglyceride, HDL-C, LDL-C) | Days 1, 28, and 56
  Blood lipid will be measured at the beginning, 4-week, and 8-week time points.
Change from baseline in blood coagulation factor (factor VII, fibrinogen) | Days 1, 28, and 56
  Blood coagulation factor will be measured at the beginning, 4-week, and 8-week time points.
Change from baseline in arteriosclerosis | Days 1 and 56
  Arteriosclerosis will be measured by B-scan ultrasonography at the beginning and 8-week time points.

SECONDARY OUTCOMES:
Change from baseline in blood glucose | Days 1, 28, and 56
  Blood glucose will be measured at the beginning, 4-week, and 8-week time points.
Change from baseline in blood hs-CRP | Days 1 and 56
  Blood hs-CRP will be measured at the beginning 8-week time points.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Fengxian District Central Hospital, Shanghai, China